CLINICAL TRIAL: NCT04144205
Title: Effect of Arterial Oxygen Partial Pressure on Mixed Venous Oxygen Saturation and Regional Cerebral Oxygen Saturation During Cardiopulmonary Bypass in Patients Undergoing Cardiac Surgery: a Pilot Study
Brief Title: Effect of Arterial Oxygen Partial Pressure on Mixed Venous Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PaO2 and SvO2
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fraction of inspired oxygen setting change (Experimental)
  Interventions: Other: Change of the fraction of inspired oxygen

INTERVENTIONS:
Other: Change of the fraction of inspired oxygen — After the stabilization of cardiopulmonary bypass, in the first half of patients, fraction of inspired oxygen would be set at 0.5 and maintained for 5 minutes (T0), then it would be changed to 1.0 and maintained for 5 minutes (T1). Again, fraction of inspired oxygen would be resumed to be 0.5 and maintained for 5 minutes (T2).
  In the other half of patients, the direction of change in fraction of inspired oxygen will be reversed as follows. It will be set at 1.0 and maintained for 5 minutes (T0), then changed to 0.5 and maintained for 5 minutes (T1), and finally to 1.0 and maintained for 5 minutes (T2).

SUMMARY:
Mixed venous oxygen saturation is known to reflect oxygen delivery and, thus, is frequently monitored in patients undergoing cardiac surgery. Factors that affect mixed venous oxygen saturation include hemoglobin level, arterial oxygen saturation and arterial oxygen partial pressure. Among them, arterial oxygen partial pressure is known to have minimal effect on oxygen delivery compared to hemoglobin and arterial oxygen saturation. However, some argues that in certain clinical setting, such as anemia which is very common in cardiac surgery patients, the contribution of plasma (arterial oxygen partial pressure in this case) to oxygen delivery becomes more significant. Therefore, we planned to perform a pilot clinical trial to observe the change of oxygen delivery, which would be reflected in mixed venous oxygen saturation and cerebral regional oxygen saturation, according to hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* Patients that scheduled to undergo cardiac surgery using cardiopulmonary bypass.

Exclusion Criteria:

* Emergent surgery
* Symptomatic carotid artery stenosis or carotid artery stenosis of ≥50%
* Preoperative oxygen therapy that is equivalent to the inspired oxygen fraction of 0.5.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Mixed venous oxygen saturation | From the beginning and the stabilization of cardiopulmonary bypass to 15 minutes thereafter.
  Change of mixed venous oxygen saturation according to the fraction of inspired oxygen

SECONDARY OUTCOMES:
Cerebral regional oxygen saturation | From the beginning and the stabilization of cardiopulmonary bypass to 15 minutes thereafter.
  Change of cerebral regional oxygen saturation according to the fraction of inspired oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea